CLINICAL TRIAL: NCT02333188
Title: A Genotype-Guided Dosing Study of FOLFIRABRAX in Previously Untreated Patients With Advanced Gastrointestinal Malignancies
Brief Title: Genetic Analysis-Guided Dosing of FOLFIRABRAX in Treating Patients With Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0595; NCI-2014-02407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-0595 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Adenocarcinoma of Unknown Primary; Adult Cholangiocarcinoma; Gallbladder Carcinoma; Gastric Adenocarcinoma; Malignant Gastrointestinal Neoplasm; Metastatic Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma; Stage III Ampulla of Vater Cancer; Stage III Pancreatic Cancer; Stage IIIA Gallbladder Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gallbladder Cancer; Stage IIIB Gastric Cancer; Stage IV Ampulla of Vater Cancer; Stage IV Gallbladder Cancer; Stage IV Gastric Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (FOLFIRABRAX) (Experimental): Patients receive FOLFIRABRAX comprising paclitaxel albumin-stabilized nanoparticle formulation IV over 0.5 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 1.5 hours, and fluorouracil IV over 46 hours on days 1 and 15. Courses repeat every 4 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Drug: Leucovorin Calcium; Drug: Irinotecan Hydrochloride; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane
Drug: Leucovorin Calcium — Given IV
  Other Names: CF
Drug: Irinotecan Hydrochloride — Given IV
Drug: Fluorouracil — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects of genetic analysis-guided dosing of paclitaxel albumin-stabilized nanoparticle formulation, fluorouracil, leucovorin calcium, and irinotecan hydrochloride (FOLFIRABRAX) in treating patients with gastrointestinal cancer that has spread to other parts of the body and usually cannot be cured or controlled with treatment. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, fluorouracil, leucovorin calcium, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Genetic analysis may help doctors determine what dose of irinotecan hydrochloride patients can tolerate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicity (DLT) rate in cycle #1 in each of three uridine diphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) genotype groups (*1/*1, *1/*28, *28/*28) using genotype-guided dosing of irinotecan (irinotecan hydrochloride) as part of the FOLFIRABRAX regimen.

SECONDARY OBJECTIVES:

I. To determine the cumulative dose of each chemotherapy drug (nab-paclitaxel [paclitaxel albumin-stabilized nanoparticle formulation], irinotecan, 5-FU [fluorouracil]) administered in each genotype group.

II. To determine the response rates (in patients with measurable disease) by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) for each different disease (pancreatic cancer, biliary tract cancer, esophageal/gastric cancer, adenocarcinoma of unknown primary) treated in the study.

OUTLINE:

Patients receive FOLFIRABRAX comprising paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 0.5 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 1.5 hours, and fluorouracil IV over 46 hours on days 1 and 15. Courses repeat every 4 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma, gastric adenocarcinoma, cholangiocarcinoma, gall bladder adenocarcinoma, ampullary carcinoma, adenocarcinoma of unclear primary (with a gastrointestinal primary suspected), or other primary gastrointestinal malignancy for which the treating physician feels that FOLFIRABRAX is a reasonable therapeutic option
* Patients with a history of obstructive jaundice due to the primary tumor must have a metal biliary stent in place
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy > 3 months
* Absolute neutrophil count (ANC) >= 1500/ul
* Hemoglobin > 9 g/dL
* Platelets > 100,000/ul
* Total bilirubin =< 1.25 times upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal
* Alkaline phosphatase =< 2.5 times the upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Creatinine =< 1.5 mg/dL
* Measurable or non-measurable disease will be allowed, but only those with measurable disease will be evaluable for the response rate endpoint
* Women of childbearing potential and sexually active males must use an effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test at screening for patients of childbearing potential
* Signed informed consent

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for any cancer
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Diarrhea, grade 1 or greater by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version [v.] 4.0); pancreatic cancer patients with clinical evidence of pancreatic insufficiency must be taking pancreatic enzyme replacement
* Neuropathy, grade 2 or greater by NCI-CTCAE, v. 4.0
* Documented brain metastases
* Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment
* Active uncontrolled bleeding
* Pregnancy or breastfeeding
* Major surgery within 4 weeks
* Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been previously treated and the lifetime recurrence risk is less than 30%
* Patients taking substrates, inhibitors and inducers of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) should be encouraged to switch to alternative drugs whenever possible
* Patients with any polymorphism in UGT1A1 other than *1 or *28 (e.g., *6)
* History of interstitial lung disease, idiopathic pulmonary fibrosis, silicosis or connective tissue disorders
* Subjects known to be human immunodeficiency virus (HIV)-positive, including those on combination antiretroviral therapy, are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
DLT rate in course 1 for each of the three genotype groups, graded according to NCI CTCAE v 4.0 | 4 weeks

SECONDARY OUTCOMES:
Incidence of adverse events graded according to NCI CTCAE v 4.0 | Up to 6 months
  Adverse events will be summarized by type, grade, and attribution.
Response rates (by RECIST 1.1) for patients with each different type of gastrointestinal malignancy | Up to 6 months
  These results will be compared descriptively to appropriate historical controls. Exact 90% confidence intervals will be generated for the response rates.
Cumulative doses of the drugs will be calculated as the sum of all doses received on protocol therapy for each patient | Up to 6 months
  The means and standard deviations for patients in each genotype group will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (8):
- United States (8):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Fort Wayne Medical Oncology/Hematology, Fort Wayne, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Virginia Mason, Seattle, Washington